CLINICAL TRIAL: NCT02532699
Title: Anti-hypertensive Effect of Fermented Mycelia of Antrodia Cinnamomea Among Mild Hypertensive Subjects in a Double-blinded Randomized Trial
Brief Title: Anti-hypertensive Effect of Mycelia of Antrodia Cinnamomea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Principal Investigator, You-Cheng Shen, School of Health Diet and Industry Managment, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CS11043; E099N0115-MY2 (Other Grant/Funding Number: Grape King Bio Ltd)
Record Dates: First submitted 2015-08-14; First posted 2015-08-26 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension
Keywords: Antrodia cinnamomea mycelia; blood pressure; adenosine; antrosterol; clinical trial; gamma-aminobutyric acid
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AC mycelia (Active Comparator): Subjects receive three capsules per day containing either 420 mg of AC mycelia.
  Interventions: Dietary Supplement: AC mycelia
- Placebo (Placebo Comparator): Subjects receive three capsules per day containing starch placebo of similar appearance.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: AC mycelia — An 8 week double-blinded randomized placebo-controlled parallel study with 2 week follow-up period was performed in mild hypertension subjects. Consenting eligible subjects were receive three capsules per day containing either 420 mg of AC mycelia of similar appearance for 8 weeks. The subjects were required to visit at baseline, every two weeks during the intervention period (8 weeks), and at follow-up 2 weeks after treatment had ended. During each study visit, systolic and diastolic BPs were recorded, fasting blood samples were collected and anthropometric measurements were performed. Compliance was evaluated using a food diary and monitored with biweekly telephone calls.
  Other Names: niu-chang-chih
  Arms: AC mycelia
Dietary Supplement: Placebo — An 8 week double-blinded randomized placebo-controlled parallel study with 2 week follow-up period was performed in mild hypertension subjects. Consenting eligible subjects were receive three capsules per day containing 420 mg starch placebo of similar appearance for 8 weeks. The subjects were required to visit at baseline, every two weeks during the intervention period (8 weeks), and at follow-up 2 weeks after treatment had ended. During each study visit, systolic and diastolic BPs were recorded, fasting blood samples were collected and anthropometric measurements were performed. Compliance was evaluated using a food diary and monitored with biweekly telephone calls.
  Arms: Placebo

SUMMARY:
This the first report undertaken to assess the effect of supplementation with oral gamma-aminobutyric acid (GABA), adenosine and antrosterol-containing AC mycelia on blood pressure among people with mild hypertension. Overall, AC mycelia consumption for 8 weeks could successfully reduce mean diastolic and systolic BP through the suppression of PRA that is linked to downstream suppresion of angiotensin II formation, which further decreases the sympathetic outflow that leads to hypertension. In addition to blood pressure lowering properties, AC mycelia also has beneficial effect in reducing oxidative stress, significantly. No adverse events were noted, suggesting that AC mycelia deserve its consideration as a candidate for safe alternative treatment to conventional anti-hypertensive medications.

DETAILED DESCRIPTION:
This the first report undertaken to assess the effect of supplementation with oral gamma-aminobutyric acid (GABA), adenosine and antrosterol-containing AC mycelia on blood pressure among people with mild hypertension. Forty-one subjects with systolic blood pressure (SBP) between 130 and 179 mm Hg and/or diastolic blood pressure (DBP) between 85 and 109 mm Hg were randomized to receive either AC mycelia or starch placebo for 8 weeks, and had follow-up observation for an additional 2 weeks. SBP in the subjects given GABA, adenosine and antrosterol-rich AC mycelia significantly decreased compared to those who received the placebo (p<0.05). DBP also decreased after the intake of AC mycelia. Compared to the placebo, AC mycelia significantly reduced plasma renin activity by a maximum of 25 % and 36 % on week 8. This suppression suggested that AC mycelia is a potent inhibitor of renin, and its bioavailability is sufficient to produce BP reduction after a short term of oral administration. Neither adverse events nor abnormal laboratory findings were noted throughout the study period, suggesting that GABA, adenosine and antrosterol-rich AC mycelia significantly decreased borderline hypertension, which may support its consideration as a safe alternative treatment compared to conventional anti-hypertensive medications.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects were untreated hypertensive men or women aged between 20 and 80 years old with SBP between 130 and 179 mmHg and/or DBP between 85 and 109 mmHg as measured in a sitting position

Exclusion Criteria:

* Subjects were excluded if they had a history of major cardiovascular disease, severe liver dysfunction, insulin-dependent diabetes mellitus or stroke. They were also excluded if they routinely consumed alcohol, were pregnant or unable to comprehend study instructions.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-06; Primary Completion 2012-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
AC anti-hypertensive measure blood pressure (SBP and DBP ) | 10 weeks
  "Blood pressure" to "Number of pressure with SBP and DBP,

SECONDARY OUTCOMES:
Blood biochemical values (Liver function) | 10 weeks
  values of liver function with AST and ALT

CONTACTS AND LOCATIONS:
Overall Officials: You-Cheng Mr Shen, Ph.D., Principal Investigator — Chung Shan Medical University

REFERENCES:
- [Background] 1. Geethangili, M.; Tzeng, Y.M. Review of pharmacological effects of antrodia camphorata and its bioactive compounds. Evidence-based complementary and alternative medicine : eCAM 2011, 2011, 212641. 2. Liu, D.Z.; Liang, Y.C.; Lin, S.Y.; Lin, Y.S.; Wu, W.C.; Hou, W.C.; Su, C.H. Antihypertensive activities of a solid-state culture of taiwanofungus camphoratus (chang-chih) in spontaneously hypertensive rats. Bioscience, biotechnology, and biochemistry 2007, 71, 23-30. 3. Jong-Wook Shin, S.-I.L.; Kim, S.-D. Effect of acetic acid fermented juice prepared using submerged culture media of antrodia camphorata mycelium on blood glucose and lipid profiles of rats in which diabetes was induced with streptozotocin. Korean J. Food Preserv. 2008, 15, 725-730.